CLINICAL TRIAL: NCT05912114
Title: Effectiveness of 1L Mannitol Versus 1L Polyethylene Glycol Electrolyte Dispersion as a Salve for Patients With Inadequate Bowel Preparation: a Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Mannitol Versus Polyethylene Glycol Electrolyte Dispersion as a Salve for Patients With Inadequate Bowel Preparation: a Randomized Controlled Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MPEG1.0
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Bowel Cleansing; Good Taste
MeSH Terms: interventions — Mannitol; glycoprep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mannitol (Experimental): Use of oral 1L Mannitol for remediation of intestinal uncleanliness
  Interventions: Drug: Mannitol
- Polyethylene glycol electrolyte (Active Comparator): Use of oral 1L PEG for remediation of intestinal uncleanliness
  Interventions: Drug: Polyethylene glycol electrolyte

INTERVENTIONS:
Drug: Mannitol — Mannitol, as an osmotic laxative, increases the colloid osmotic pressure in the intestinal lumen, which results in a hyperosmolar state in the intestine, thus allowing easy elimination of stools.
  Arms: Mannitol
Drug: Polyethylene glycol electrolyte — Polyethylene glycol electrolyte is an inert polymer that cannot be absorbed by the body itself. Due to its high permeability, it retains water in the intestinal tract, increasing the amount of fluid retained in the intestine and softening the stool, thus acting as a diuretic.
  Arms: Polyethylene glycol electrolyte

SUMMARY:
For patients with inadequate bowel preparation, current guidelines recommend either remedial measures or rescheduling the endoscopy, but previous surveys have found that approximately 30% of patients do not follow medical advice to reschedule the examination if it is rescheduled, while those who take remedial measures on the same day are more compliant, so remedial measures may be a better option than rescheduling the examination. As for the remedy regimen, it has been demonstrated that oral PEG is superior to the enema regimen in terms of bowel cleansing, but PEG is very resistant to be taken by most patients due to its poor taste and the larger doses required, resulting in poor bowel preparation and poor compliance. In contrast, oral mannitol has the advantages of small dose and good taste, and patient compliance may be higher.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years with a pre-first colonoscopy bowel cleanliness of less than 2 points in any segment of the bowel.

Exclusion Criteria:

- (1) Pregnant women. (2) History of colorectal surgery. (3) Patients with acute exacerbation of inflammatory bowel disease. (4) Patients with severe medical conditions that make them unsuitable for colonoscopy.

(5) Patients with known allergy to mannitol/PEG. (6) Patients who refuse to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Bowel cleanliness | 1 hour
  The BBPS scoring method, defined as a score of ≥2 for each bowel segment, was used to consider the preparation adequate.

SECONDARY OUTCOMES:
Patients' feelings | 1 hour
  Patients' perceptions of the taste and ease of use of the two drugs.

OTHER OUTCOMES:
Patients' willingness to take such measures again. | 1 hour
  Patient's willingness to take the same medication before the next colonoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China

REFERENCES:
- [Derived] Zheng S, Xu Z, Deng F, Wang S, Qian T, Lin P, Wang C, Wang W, Xia Y, Xu L, Zhang Z. Comparing the efficacy of mannitol and polyethylene glycol in treating patients with poor bowel preparation: a randomized controlled clinical study. Tech Coloproctol. 2025 Dec 24;30(1):15. doi: 10.1007/s10151-025-03243-y. PMID 41444456